CLINICAL TRIAL: NCT03289494
Title: A Pilot Randomized Controlled Trial Evaluating the Effect of Two Diets With Different Starch Digestibility Profiles on Daily Glycemic Profile Measured by Continuous Glucose Monitoring System (CGMS), in Type 2 Diabetic Patients
Brief Title: Evaluation of 2 Diets With Different Starch Digestibility Profiles on Daily Glycemic Profile, in T2D Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other); Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KBE052
Record Dates: First submitted 2017-09-13; First posted 2017-09-21 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Type2 Diabetes
Keywords: Slowly Digestible Starch; SDS; Type 2 diabetes; T2D; Glycemic response; Continuous Glucose Monitoring System; CGMS
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Each subject will receive two independant weeks of diet intervention, in a crossover design
Who Masked: Participant
Masking Description: Each diet will be labelled "Diet A" or "Diet B"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet A (Active Comparator): Balanced diet high in Slowly Digestible Starch
  Interventions: Other: Balanced diet high in Slowly Digestible Starch
- Diet B (Placebo Comparator): Balanced diet low in Slowly Digestible Starch
  Interventions: Other: Balanced diet low in Slowly Digestible Starch

INTERVENTIONS:
Other: Balanced diet high in Slowly Digestible Starch — The carbohydrate present in the diet high in Slowly Digestible Starch were selected according to the general recommendations made for diabetics and according to their SDS content. The diet will be consumed during one week.
  Arms: Diet A
Other: Balanced diet low in Slowly Digestible Starch — The carbohydrate present in the diet low in Slowly Digestible Starch were selected according to the general recommendations made for diabetics and according to their SDS content. The diet will be consumed during one week.
  Arms: Diet B

SUMMARY:
The study is a randomized cross-over pilot study. The research hypothesis is that the diet high in SDS content (H-SDS) will lower the daylong glycemic response and improve the glycemic control in patients with type 2 diabetes (T2D) compared to the diet low in SDS content (L-SDS).

DETAILED DESCRIPTION:
The study is a randomized cross-over pilot study. The research hypothesis is that the diet high in SDS content (H-SDS) will lower the daylong glycemic response and improve the glycemic control in patients with type 2 diabetes (T2D) compared to the diet low in SDS content (L-SDS).

8 patients with type 2 diabetic patients will be recruited.

Subjets will have 5 visits:

The selection visit (V1) is required to check whether the patients fulfill inclusion and exclusion criteria for the study.

The visit V2 will include randomization, medical check-up and a dietary interview (LogBook supply with explanations for filling and dietary advice cards for the 1st week of diet). The nurse will insert the CGMS and the patient will receive detailed instructions on wearing the sensor and recorder. The patient will leave the research center with a glucometer, the starchy foods and cereal products adapted for its first week of diet and the associated cooking instruction sheets and menus given by the dietician.

During each day of the first experimental diet period, the patient will take at least four blood glucometer readings per day, and will consume the food products according to a menu plan and the cooking instruction sheets given by the dietician, and fill a dietary record.

After 6 days +/- 1 day, the patient will return to the center (Visit V3) to remove the CGMS, bring back the glucometer and the follow-up LogBook. A Medical check-up will also be performed. Compliance will be assessed using the dietary record of the follow-up LogBook and the return of the uneaten products (weighting). A feedback questionnaire will be completed by each patient to have a global assessment of the diet and to evaluate the feasibility of this type of diet over longer periods.

The wash-out period will then last 2 weeks +/- 3 days. Then a new sequence will start. The visit V4 will be similar to visit V2 with: installation of the CGMS, provision of the LogBook and diet specific information for the second period. The glucometer and starchy foods and cereal products will be supplied to the patients.

During each day of this second diet period, patients will be required to consume starchy foods and cereal products according to a menu plan and cooking instructions provided by the dietician, and fill a dietary record. The patient will realize 4 capillary blood glucose control and will fill the information required in the LogBook.

Finally, Visit V5 will be the last visit. It will include, like for visit V3: removal of CGMS, return of glucometer and follow-up LogBook and a medical check-up . Compliance will be assessed using the dietary record of the follow-up LogBook and the return of the uneaten products (weighting). A feedback questionnaire will be completed by patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient able to understand the study information and providing written consents for his/her participation to the study
* Male or female
* Patient undergoing medical examination during the selection visit
* Patient aged between 18 and 75 years old (bounds included)
* T2D volunteer with:

  * HbA1c between 6,5% and 8,5%
  * Bi-therapy associating metformin and sitagliptin at stable dose for at least 1 month
* T2D volunteer without insulin therapy or GLP-1 analogues
* Patient with BMI ranging between 22 and 37 kg/m2 (bounds included)
* Patient with stable body weight over the past three months (+/- 5 % of body weight)
* Patient accepting to change its diet for two weeks
* Patient not suffering from intolerance or allergy
* Patient regularly consuming products proposed in the study
* Patient regularly consuming 3 main meals per day
* Sedentary behavior or stable regular physical activity during the study
* Patient not presenting any disease during the medical examination / interview which could interfere with the results of the study according to the investigator
* Patient covered by health assurance

Exclusion Criteria:

* General criteria:

  * Patient under legal protection measure
  * Patient deprived of liberty by a court or an administrative decision
  * Patient currently participating in another study or being in the exclusion period of another study
  * Volunteer that exceed the financial compensation allowed per year for participating in research programs
* Biological criteria:

  * Gamma-GT > 2.5 times above the norm (>160 UI/L)
  * ASAT > 2.5 times above the norm (>85 UI/L)
  * ALAT > 2.5 times above the norm (>137.5 UI/L)
  * Triglycerides > 4 g/L
  * LDL-cholesterol > 1.90 g/L
  * CRP > 15 mg/L
  * Hemoglobin < 120 mg/dL
  * Other biological abnormality with clinical significant relevance according to the investigator
* Therapeutic and medical criteria:

  * Patient with type 1 diabetes
  * T2D treatment other than metformin and sitagliptin
  * Patient with past bariatric surgery
  * Patient with medical history of endocrine diseases who may interfere with glucose metabolism according to the investigator (such as thyroid dysfunction, acromegaly, hypercorticism…)
  * Uncontrolled high blood pressure defined by Systolic blood pressure > 150 mmHg or Diastolic blood pressure > 100 mmHg
  * Evidence of any other unstable or untreated clinically significant immunological, neoplasic, endocrine, haematological, gastrointestinal, hepatic, neurological or psychiatric abnormalities or medical disease according to the investigator
  * Pregnant women or willing to become pregnant or lactating women
  * Women of childbearing age without an efficient contraceptive method according to the investigator
  * Patient under a restrictive diet or willing to lose weight
  * Patient with eating disorders (e.g. anorexia nervosa and bulimia) according to the investigator
  * Patient without stable dietary habits or with specific diet (vegetarian, vegan,…) according to the investigator
  * Patient who smokes
  * Patient regularly consuming more than 20 g/day of alcohol. Consumption of more than 3 alcoholic beverages per day is recognized as excessive. An alcoholic beverage is: 30 mL of spirituous, 120 mL of wine or 330 mL of beer
  * Patient regularly consuming recreational drugs
  * Patient consuming in the two previous months regularly corticoids, anorectics, adrenergic drugs, beta-blocking drugs, antiplatelet agent (like aspirin) or other drugs or supplement that should impact glucose metabolism (other than metformin or DPP4 inhibitor) in the investigator's opinion
  * Adhesive plaster skin allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Mean postprandial incremental Area Under the Curve (iAUC), measured by CGMS | minimum 2h to maximum 6h postprandial periods and average value of minimum 3 days to a maximum of 6 days of CGMS record
  The iAUC will be calculated using the trapezoid rule. The iAUC includes all area below the curve and above the fasting concentration, with any area beneath fasting being ignored.

SECONDARY OUTCOMES:
Glycemic profile parameters: Minimum glycaemia | minimum 3 days to a maximum of 6 days of CGMS record
  Minimum glycaemia
Glycemic profile parameters: maximum glycaemia | minimum 3 days to a maximum of 6 days of CGMS record
  maximum glycaemia
Glycemic profile parameters: Standard Deviation (SD) from CGMS glycaemia | minimum 3 days to a maximum of 6 days of CGMS record
  Standard Deviation (SD) from CGMS glycaemia
Glycemic profile parameters: Coefficient of Variation (CV) from CGMS glycaemia | minimum 3 days to a maximum of 6 days of CGMS record
  Coefficient of Variation (CV) from CGMS glycaemia
Glycemic profile parameters: MAGE | minimum 3 days to a maximum of 6 days of CGMS record
  Mean Amplitude of Glycemic Excursions (MAGE) from CGMS glycaemia
Glycemic profile parameters: MODDs | minimum 3 days to a maximum of 6 days of CGMS record
  Mean Of Daily Differences (MODDs) from CGMS glycaemia
Glycemic profile parameters: MIME | minimum 3 days to a maximum of 6 days of CGMS record
  Mean Indices of Meal Excursions (MIME) from CGMS glycaemia
Glycemic profile parameters: Time in Range | minimum 3 days to a maximum of 6 days of CGMS record
  Mean time spent in the appropriate glycemic range in %
Glycemic profile parameters: ADRR | minimum 3 days to a maximum of 6 days of CGMS record
  Average of Daily Risk Ratio (ADRR) from CGMS glycaemia
Glycemic profile parameters: CONGA | minimum 3 days to a maximum of 6 days of CGMS record
  Continuous Overall Net Glycemic Action (CONGA) from CGMS glycaemia
Glycemic profile parameters: hyperglycemia durations | minimum 3 days to a maximum of 6 days of CGMS record
  hyperglycemia durations
Glycemic profile parameters: hypoglycemia durations | minimum 3 days to a maximum of 6 days of CGMS record
  hypoglycemia durations
Glycemic profile parameters: mean glycemic value | minimum 3 days to a maximum of 6 days of CGMS record
  mean glycemic value on relevant time interval
Glycemic profile parameters: incremental AUC | minimum 3 days to a maximum of 6 days of CGMS record
  incremental AUC calculated on relevant time interval
Glycemic profile parameters: total AUC | minimum 3 days to a maximum of 6 days of CGMS record
  total AUC calculated on relevant time interval, calculated using the trapezoid rule and including all area below the curve
Glycemic profile parameters: kinetics | minimum 3 days to a maximum of 6 days of CGMS record
  Daylong glycaemia kinetics
Compliance parameters: mean SDS ingestion | maximum of 6 days of LogBook record
  mean SDS ingestion by type of meal and per day
Dietary intake evaluation | After 1 week intervention diet
  Dietary record analysis, in g of macronutrient intake
Dietary record evaluation | After 1 week intervention diet
  Dietary record analysis, in % of total energy intake
Charaterisation of acceptability to H-SDS diet in free living conditions | After 1 week intervention diet
  Feedback questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DISSE, MD, PhD, Principal Investigator — Centre de Recherche en Nutrition Humaine Rhône-Alpes; Martine LAVILLE, MD, PhD, Study Chair — Centre de Recherche en Nutrition Humaine Rhône-Alpes
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhone-Alpe, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breyton AE, Goux A, Lambert-Porcheron S, Meynier A, Sothier M, VanDenBerghe L, Brack O, Disse E, Laville M, Vinoy S, Nazare JA. Starch digestibility modulation significantly improves glycemic variability in type 2 diabetic subjects: A pilot study. Nutr Metab Cardiovasc Dis. 2021 Jan 4;31(1):237-246. doi: 10.1016/j.numecd.2020.08.010. Epub 2020 Aug 25. PMID 32988721